CLINICAL TRIAL: NCT02941744
Title: A Phase IB Clinical Trial on Adjuvant Low-dose Ipilimumab Plus Nivolumab Following the Resection of Melanoma Macrometastases
Brief Title: A Clinical Trial: Adjuvant Low-dose Ipilimumab + Nivolumab After Resection of Melanoma Macrometastases
Acronym: ipniv
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-BN-001
Record Dates: First submitted 2016-09-14; First posted 2016-10-21 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
Keywords: nivolumab; ipilimumab; low fixed dose; adjuvant therapy; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IpNiv (Experimental): low fixed dose ipilimumab plus low fixed dose nivolumab
  Interventions: Drug: nivolumab; Drug: ipilimumab

INTERVENTIONS:
Drug: nivolumab — low fixed dose ipilimumab in combination with nivolumab
  Other Names: Opdivo
Drug: ipilimumab — low fixed dose ipilimumab in combination with nivolumab
  Other Names: Yervoy

SUMMARY:
Nivolumab (OpdivoTM, BMS), a human IgG-4 anti-PD-1 monoclonal antibody has demonstrated anti-tumor activity in patients with advanced melanoma.

The investigators postulate that patients with melanoma nivolumab have a comparable tumor response rate at a dose range of 0.1 to 10 mg/kg q2wks.

Ipilimumab (YervoyTM, BMS), a human IgG-1 anti-CTLA-4 monoclonal antibody improves the survival of patients with advanced melanoma. Adjuvant therapy with ipilimumab improves the relapse-free survival after complete resection of high-risk stage III melanoma (EORTC 18071).

Combined treatment with ipilimumab plus nivolumab improves the tumor response rate and overall survival of patients with advanced melanoma but is associated with a higher incidence of immune related adverse events (CheckMate 067).Nivolumab and ipilimumab have distinct immunological mechanisms that can be revealed by analyzing TCR usage in blood lymphocytes.

DETAILED DESCRIPTION:
Currently, there is no standard of care or no available treatment for subjects with AJCC Stage IIIb/c and Stage IV NED melanoma who are at high risk for recurrence following complete resection of their metastasis. Ipilimumab (10mg/kg), interferon, pegylated interferon therapy or observations alone are the typical options for the Stage III patients who achieve a complete resection and are Food and Drug Administration (FDA) approved. In the EU, high-dose interferon is the only approved drug for the adjuvant treatment of melanoma patients. Given the unexceptional benefit and high toxicity profile in a patient population that is free of disease, it is controversial whether ipilimumab and interferon can be considered standard of care for Stage III melanoma. Nivolumab, a PD1 blocking monoclonal antibody, has shown superior anti-tumor activity across a wide range of dose-levels (0,1 to 10 mg/kg every 2 weeks) in patients with advanced melanoma. Nivolumab (at a dose of 3 mg/kg every 3 weeks) demonstrated a survival benefit in treatment naive patients with BRAF Wild Type (WT), metastatic melanoma in a Phase 3, randomized clinical trial and a PFS benefit over ipilimumab as a first-line therapy for advanced melanoma. Combination therapy with ipilimumab and nivolumab results in a higher response rate and PFS as compared to the results obtained with monotherapy. Combination therapy however significantly increases the incidence of grade > 3 adverse events, to the extent that this regimen would probably be associated with unacceptable toxicity in the adjuvant setting. The toxicity seems to be driven by Ipilimumab. The adverse events seen on Ipilimumab are dose dependent.

Unlike PD-1 blockade, CTLA-4 blockade diversifies the peripheral T-cell pool, representing a pharmacodynamic effect that can be measured by a DNA-sequencing technology referred to as ImmunoSeq.

This phase IB study will investigate the effect of low-dose ipilimumab and low-dose nivolumab on the peripheral T-cell repertoire of patients who are free of disease following the resection of melanoma macrometastases.

Treatment with low-dose ipilimumab in combination with low-dose nivolumab will be safe and modify the peripheral T-cell repertoire in subjects with completely resected Stage IIIb/c and Stage IV melanoma who are at high risk for recurrence.

Ipilimumab (YervoyTM, BMS), a human IgG-1 anti-CTLA-4 monoclonal antibody improves the survival of patients with advanced melanoma .Adjuvant therapy with ipilimumab improves the relapse-free survival after complete resection of high-risk stage III melanoma .

Combined treatment with ipilimumab plus nivolumab improves the tumor response rate and overall survival of patients with advanced melanoma but is associated with a higher incidence of immune related adverse events.

Nivolumab and ipilimumab have distinct immunological mechanisms that can be revealed by analyzing TCR usage in blood lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be either Stage IIIb/c or Stage IV AJCC (7th edition) and have histologically confirmed melanoma that is completely surgically resected in order to be eligible. Subjects must have been surgically rendered free of disease with negative margins on resected specimens. Please refer to Appendix 1 or description of AJCC 7th editions of TNM and staging.
* If Stage III melanoma (whether Stage IIIb or IIIc) the subjects must have clinically detectable lymph nodes that are confirmed as malignant on the pathology report Clinically detectable lymph nodes are defined as:

  * A palpable node (confirmed as malignant by pathology)
  * A non-palpable but enlarged lymph node by CT (at least 15 mm in short axis) and confirmed as malignant by pathology
  * A PET positive lymph node of any size confirmed by pathology
  * Evidence of pathologically macrometastatic disease in one or more lymph nodes defined by one or more foci of melanoma at least 1cm in diameter

    * All melanomas, except ocular/uveal melanoma, regardless of primary site of disease will be allowed
    * Complete resection of Stage III disease that is documented on the surgical and pathology reports or complete resection of Stage IV disease with margins negative that is documented on the pathology report.
    * Complete resection must be performed within 16 weeks prior to recruitment
    * Subjects must not have received systemic medical anti-cancer treatment (postsurgical local/locoregional radiation therapy applied according to local standard practice is allowed)
    * All subjects must have disease-free status documented by a complete physical examination and total body PET/CT imaging within 4 weeks prior to recruitment.
    * ECOG performance status score of 0 or 1 (Appendix 2)
    * In order to be recruited, tumor tissue from the resected site of disease must be provided for biomarker analyses. If insufficient tumor tissue content is provided for analysis, acquisition of additional archived tumor tissue (block and /or slides) for the biomarker analysis is required.
    * Prior treated central nervous system (CNS) metastases must be without MRI evidence of recurrence for at least 4 weeks after treatment, subjects must be off immunosuppressive doses of systemic steroids (> 10 mg/day or equivalent) for at least 14 days prior to study drug administration, and must have returned to neurologic baseline post-operatively. The 4-week period of stability is measured after the completion of the neurologic interventions, ie surgery and/or radiation
    * In addition to neurosurgery to treat CNS metastases, adjuvant radiation after the resection of CNS metastasis is allowed. Immunosuppressive doses of systemic steroids (doses < 10 mg/day prednisone or equivalent) must be discontinued at least 14 days before study drug administration
    * Prior surgery that required general anesthesia must be completed at least 4 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration.
    * All baseline laboratory requirements will be assessed and should be obtained within 14 days of recruitment. Screening laboratory values must meet the following criteria:

      i. WBCs > 2000/μL ii. Neutrophils > 1500/μL iii. Lymphocytes > 1000/μL iv. Platelets > 100 x 10³/μL v. Hemoglobin > 9.0 g/dL vi. Creatinine Serum creatinine <1.5 x upper limit of normal (ULN) or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula) vii. AST < ULN viii. ALT < ULN ix. Total Bilirubin < 1 x ULN (except subjects with Gilbert Syndrome who must have total bilirubin < 3.0 mg/dL) x. LDH < 1,5x ULN xi. CRP < 2x ULN

Exclusion Criteria:

* Subjects with leptomeningeal metastases
* History of ocular/uveal melanoma
* Medical History and Concurrent Diseases

  * Subjects with previous non-melanoma malignancies are excluded unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required or anticipated to be required during the study period (exceptions include but are not limited to, non-melanoma skin cancers; in situ bladder cancer, in situ gastric cancer, or in situ colon cancers; in situ cervical cancers/dysplasia; or breast carcinoma in situ)
  * Subjects with active, known, or suspected autoimmune disease. Subjects with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that a BMS medical monitor be consulted prior to signing informed consent.
  * Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
  * Prior therapy for melanoma except surgery for the melanoma lesion(s) and except adjuvant RT after neurosurgical resection for CNS lesions. Specifically subjects who received prior therapy with interferon, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways) are not eligible.
  * Treatment directed against the resected melanoma (eg, chemotherapy, targeted agents, biotherapy, or limb perfusion) that is administered after the complete resection.
  * Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive protocol therapy.
* Physical and Laboratory Test Findings

  * Positive test for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection.
  * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Allergies and Adverse Drug Reaction

  * History of Grade ≥3 allergy to humanized monoclonal antibodies
* Other Exclusion Criteria

  * Prisoners or subjects who are involuntarily incarcerated
  * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
  * Pregnant or nursing women
  * Psychological, familial, sociological, or geographical conditions that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-03; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2year
  to evaluate the safety of the investigational regimen of adjuvant low-dose ipilimumab plus nivolumab

SECONDARY OUTCOMES:
to measure t cell repertoire before and after treatment with low dose ipilimumab and nivolumab with immunoseq. | 2years
  to evaluate the effect of the investigational regimen of adjuvant low-dose ipilimumab plus nivolumab on the T-cell repertoire in the blood of subjects with completely resected Stage IIIb/c or Stage IV NED melanoma who are at high risk for recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, MD Phd, Principal Investigator — physician
Locations (1):
- UZ Brussel, Jette, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
data wil be published in total and anonymous